CLINICAL TRIAL: NCT01263366
Title: Exploratory Study of Topical Norepinephrine in Post-Surgical Breast Cancer Patients Receiving Radiotherapy
Brief Title: Exploratory Study of Norepinephrine to Prevent Radiodermatitis in Breast Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment issues
Sponsor: ProCertus BioPharm, Inc (Industry)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PC-4
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Radiodermatitis
Keywords: Radiodermatitis; Prevention; Radiotherapy; Breast; Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Norepinephrine (Experimental)
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Approximately 1.6 or 4.6 mL of a 400 mM norepinephrine solution will be applied topically to a portion of the radiation treatment field prior to each radiation treatment (20-33 treatments)
  Other Names: Noradrenaline

SUMMARY:
This study, a nonrandomized open-label Phase I safety and exploratory study, will evaluate the safety of topical norepinephrine in post-surgical breast cancer patients who are undergoing radiation therapy.

The study will also provide information about whether topical norepinephrine can prevent or decrease the severity of the radiation dermatitis experienced by these patients.

ELIGIBILITY:
Eligibility Criteria

Subjects must:

* be ≥ age 18 years of age with a documented pathological diagnosis of Stage Ia (T1, N0, M0), Stage Ib (T0 or 1, N1mic, M0) or Stage IIa (T<3cm, N0, M0) infiltrating ductal or lobular carcinoma of the breast or ductal carcinoma in situ (DCIS).
* be post-surgical patients scheduled to be treated with at least 40 to 50.4 Gy to the whole breast and axilla using either standard or hypofractionated radiation techniques . An additional 10-16 Gy boost to the lumpectomy region may also be delivered. All radiation treatment is to be delivered based on standard CT planning.
* have the ability to understand the informed consent document.
* be able to comply with protocol schedule.
* have a negative serum pregnancy test (within 7 days prior to starting radiation therapy), if a female of child bearing potential.
* consent to utilize medically acceptable methods of contraception throughout the study period if of child-bearing potential.

Exclusion Criteria

Subjects:

* with unhealed surgical wounds or scars in the study treatment area (axilla).
* with underlying active untreated cardiac disease (e.g. arrhythmia).
* with generalized skin disorders that have required treatment within the past 6 months.
* with connective tissue disorders.
* with rashes, ulcerations, or poorly healed scars in the study drug application area (axilla).
* with a known allergy to norepinephrine.
* with known uncontrolled hypertension (repeatedly elevated BP; systolic BP >139 or diastolic BP >89).
* with a known clinically significant abnormal ECG within the past 6 months.
* receiving MAO inhibitors or antidepressants (triptyline or imipramine types).
* who are pregnant or breastfeeding.
* with lymphovascular space invasion on pathology.
* with dermal lymphatic invasion on pathology.
* with proximity of the tumor to the overlying skin as evidenced by a distance of less than 5 mm on US or MRI (if performed) and within 2 cm of the anticipated application field
* diagnosis of inflammatory breast cancer.
* receiving chemotherapy other than Herceptin concurrent with the radiation.
* with previous radiation to the breast to be treated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety of daily topical application of norepinephrine to the radiation field | Safety will be assessed during the study (5-7 weeks) and at follow-up visits approximately 1, 2 and 4 weeks after the end of the treatment period.
  The primary safety hypothesis is that there will be little or no skin irritation associated with the application of the topical norepinephrine and no systemic effects secondary to transdermal absorption.

SECONDARY OUTCOMES:
Efficacy of daily topical application of norepinephrine to the radiation field | Efficacy will be assessed during the study (5-7 weeks) and at follow-up visits approximately 1, 2 and 4 weeks after the end of the treatment period.
  The primary efficacy hypothesis is that the portion of the radiation site that is treated with topical norepinephrine immediately prior to daily radiotherapy will have less severe radiation dermatitis than the adjacent untreated portion of the radiation site.

CONTACTS AND LOCATIONS:
Overall Officials: James F Cleary, MBBS, Principal Investigator — University of Wisconsin, Madison; Bethany M Anderson, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Cleary JF, Anderson BM, Eickhoff JC, Khuntia D, Fahl WE. Significant suppression of radiation dermatitis in breast cancer patients using a topically applied adrenergic vasoconstrictor. Radiat Oncol. 2017 Dec 22;12(1):201. doi: 10.1186/s13014-017-0940-7. PMID 29273054